CLINICAL TRIAL: NCT04569422
Title: Influence of Obuvacaine Hydrochloride Eye Drops on the Comfort of Meibomian Gland Massage Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Principal Investigator, JJiang Junyi, Influence of Obuvacaine Hydrochloride Eye Drops on the Comfort of Meibomian Gland Massage Patients, Aier School of Ophthalmology, Central South University
Other Study IDs: 2020-002-01
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Meibomian Gland Massage is Important to Delay the Development of Meibomian Gland Dysfunction
MeSH Terms: interventions — Benzoyl Peroxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ephedrine drop
  Interventions: Drug: Benoxyl

INTERVENTIONS:
Drug: Benoxyl — reduce pain

SUMMARY:
In this study, there were differences in patients' demands for ephedrine during meibomian gland massage and whether it would affect patients' poor comfort. Therefore, we needed to collect patients' pain grades during meibomian gland massage

DETAILED DESCRIPTION:
Meibomian gland dysfunction is a common eye disease that may be asymptomatic or painful and itchy in the early stages, requiring early daily care and medication. And meibomian gland massage is a very important step in the treatment. Meibomian gland massage is massaging along the direction of meibomian gland drainage to push out secretions that cannot be discharged by themselves, improve meibomian gland function, and delay the development of meibomian gland dysfunction.Meibomian gland dysfunction is a common eye disease that may be asymptomatic or painful and itchy in the early stages, requiring early daily care and medication. And meibomian gland massage is a very important step in the treatment. Meibomian gland massage is massaging along the direction of meibomian gland drainage to push out secretions that cannot be discharged by themselves, improve meibomian gland function, and delay the development of meibomian gland dysfunction.Meibomian gland dysfunction is a common eye disease that may be asymptomatic or painful and itchy in the early stages, requiring early daily care and medication. And meibomian gland massage is a very important step in the treatment. Meibomian gland massage is massaging along the direction of meibomian gland drainage to push out secretions that cannot be discharged by themselves, improve meibomian gland function, and delay the development of meibomian gland dysfunction.

Methods: We selected dry eye patients who visited dry eye clinic of Aier Eye Hospital from June 2020 to March 2021 to conduct questionnaire survey and analysis with pain scaleMethods: We selected dry eye patients who visited dry eye clinic of Aier Eye Hospital from June 2020 to March 2021 to conduct questionnaire survey and analysis with pain scale Group: Divided into ephedrine drop group and artificial tear drop group Research tool: Pain rating scale

ELIGIBILITY:
Inclusion Criteria:

Healthy people with no chronic disease

Exclusion Criteria:

People with chronic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Meibomian gland dysfunction people with no chronic disease
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-21 (Estimated); Study Completion 2021-05-21 (Estimated)

PRIMARY OUTCOMES:
Undifferrentiated | 2020.01-2020.09
  There was no difference in the effect of obuvacaine hydrochloride on the comfort of meibomian gland massage patients

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Yin, bachelor, Principal Investigator — Shanghai Aier Eye Hospital
Locations (1):
- Aier School of Ophthalmology, Central South University, Changsha, Hunan, China